CLINICAL TRIAL: NCT00267046
Title: A Phase II Study to Evaluate the Pharmacokinetics, Safety, and Obtain a Preliminary Efficacy Assessment of Palifermin in Patients With Sarcoma Receiving Multicycle Chemotherapy With Doxorubicin and Ifosfamide
Brief Title: Evaluate PKs and Efficacy Assessment of Palifermin in Patients With Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2004-0511
Record Dates: First submitted 2005-12-19; First posted 2005-12-20 (Estimated); Results first posted 2012-05-16 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-04

CONDITIONS: Sarcoma; Oral Mucositis
Keywords: Sarcoma; Soft Tissue Sarcoma; Oral Mucositis; Doxorubicin; Adriamycin; Ifosfamide; Palifermin; Vincristine; Cisplatin; Placebo
MeSH Terms: conditions — Sarcoma; Stomatitis | interventions — Fibroblast Growth Factor 7; Doxorubicin; Ifosfamide; Vincristine; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Palifermin (Experimental): Palifermin + Chemotherapy (Adriamycin (Doxorubicin)+ Ifosfamide (AI) or Adriamycin (Doxorubicin) + Cisplatin (AP) Regimen); Palifermin 180 mcg/kg 3 days prior to chemotherapy; Adriamycin 30 mg/m^2 intravenous (IV) for 72 hours starting Days 0 for total 90 mg/m^2. Ifosfamide 2.5 g/m^2 IV bolus Days 0-3 (total 10 g/m^2); Vincristine 2 mg IV Day 0.
  AP=Doxorubicin (Adriamycin) + Cisplatin:
  Palifermin 180 mcg/kg 3 days prior to chemotherapy; Adriamycin 30 mg/m^2 IV continuous infusion for 72 hours starting Day 0(total = 90 mg/m^2); Cisplatin 120 mg/m^2 on day 0.
  Interventions: Drug: Palifermin; Drug: Adriamycin (Doxorubicin); Drug: Ifosfamide; Drug: Vincristine; Drug: Cisplatin
- Placebo (Placebo Comparator): Placebo + Chemotherapy (AI or AP Regimen);
  AI = Doxorubicin (Adriamycin) + Ifosfamide:
  A single dose placebo prior to chemotherapy; Adriamycin 30 mg/m^2 intravenous (IV) for 72 hours starting Days 0 for total 90 mg/m^2. Ifosfamide 2.5 g/m^2 IV bolus Days 0-3 (total 10 g/m^2); Vincristine 2 mg IV Day 0.
  AP=Doxorubicin (Adriamycin) + Cisplatin:
  A single dose placebo 3 days prior to chemotherapy; Adriamycin 30 mg/m^2 IV continuous infusion for 72 hours starting Day 0(total = 90 mg/m^2); Cisplatin 120 mg/m^2 on day 0.
  Interventions: Drug: Placebo; Drug: Adriamycin (Doxorubicin); Drug: Ifosfamide; Drug: Vincristine; Drug: Cisplatin

INTERVENTIONS:
Drug: Palifermin — 180 mcg/kg 3 days prior to chemotherapy
  Arms: Palifermin
Drug: Placebo — Single dose 3 days prior to chemotherapy
  Arms: Placebo
Drug: Adriamycin (Doxorubicin) — 30 mg/m^2 IV continuous infusion for 72 hours; days 0, 1, 2 (infusion completing on day 3) (total dose = 90 mg/m^2).
  Other Names: Adriamycin
Drug: Ifosfamide — 2.5 g/m^2 IV bolus over 3 hours, days 0,1, 2, 3 (total dose = 10 g/m^2); for patients receiving the AI Regimen.
Drug: Vincristine — 2 mg IV on day 0, for patients with small cell histology receiving the AI Regimen.
Drug: Cisplatin — 120 mg/m^2 on day 0, for patients receiving the AP Regimen.
  Other Names: CDDP; Platinol

SUMMARY:
Primary:

1. To evaluate the preliminary efficacy of palifermin in reducing the incidence and severity of oral mucositis (OM) in patients with sarcoma receiving multicycle chemotherapy.
2. To evaluate the pharmacokinetics (PK) of palifermin when given pre chemotherapy.
3. To evaluate the safety profile of palifermin when combined with multicycle chemotherapy.

Exploratory:

1. To evaluate the biologic effect of palifermin on oral mucosa.
2. To investigate potential biomarker development by biochemical analysis in blood cells, serum, and plasma.
3. To investigate the effects of genetic variation in mucositis genes, drug metabolism genes, and drug target genes on patient response to the treatment regimen.

DETAILED DESCRIPTION:
Palifermin is similar to a protein keratinocyte growth factor (KGF) that is naturally made in your body in small amounts. The function of palifermin is to stimulate the growth of specific cells that form the tissue lining of your mouth and digestive tract. Damage to these cells results in the breakdown of the normal protective barrier that these cells usually provide, potentially resulting in infection.

If you are eligible to take part in this study, you will be randomly assigned (as in the toss of a coin) to receive either palifermin or placebo by vein 3 days before each cycle of chemotherapy. This will be done for 18 weeks (a total of 12 injections). A placebo is a substance that looks like the study drug, but which has no active ingredients. The infusion time will last 15-30 seconds. At the beginning of the study, for every 3 patients who are enrolled on this study, 2 of the 3 will receive palifermin. Neither you nor the study doctor will know which study drug you are assigned to receive.

Within 1 or 2 days before you receive your first dose of palifermin and between 48 to 72 hours after you receive your first dose of palifermin, additional non-invasive optical imaging procedures may be performed. The purpose of these imaging procedures is to evaluate the effects of palifermin on mucosa (mucosal thickness). The types of optical imaging that may be done include optical coherence tomography (OCT), fluorescence and reflectance spectroscopy, or confocal microscopy. The oral cavity will be inspected and photographed. A probe about the size of a pen will be placed on one or two sites of oral buccal mucosa. A beam of light will then be directed to the oral tissue and optical signals will be collected from each site. This will take about 1 minute for each site. Before using the probe for each new participant, it will be disinfected per standard practice.

You will receive adriamycin with ifosfamide or cisplatin chemotherapy. Adriamycin will be given as a continuous infusion through your central venous catheter (CVC) for 3 days. Ifosfamide will be given intravenously (intravenously (IV)--through a needle in your vein) through your CVC over 3 hours, every day for 4 days. Mesna will be given as a 24-hour IV infusion through your CVC every day for 4 days through the same catheter. Mesna is used to protect against bladder-related side effects. For patients with certain types of sarcoma, vincristine will be given through the catheter by rapid infusion on Day 1 only. In patients with bone sarcoma, cisplatin will be given on the first day as IV or intra-arterial infusion over around 4 hours instead of ifosfamide.

You will need to come in to M. D. Anderson every 3 weeks for about 4 to 5 months during the treatment period, unless your doctor decides you need to come in more frequently. At these visits, you will have your vital signs measured and routine blood tests (about 3 teaspoons each) will be performed. In addition, you may have your oral cavity examined and photographed before and after receiving the study drug. Every effort will be made to take photographs in which you cannot be identified.

Additional blood samples (about 3 teaspoons) will be taken before each cycle and as frequently as needed to measure your blood count and other tests to monitor the drug side effects and treatment effects. By the end of the study, you will have given about 10 tablespoons of blood. This amount includes the optional blood draws should you choose to allow it to be drawn.

You will be responsible for notifying study staff (at your doctors visits or over the phone with the study staff) of any side effects you experience or medications (over the counter or prescription) that you take during the treatment period. You will also be required to notify any other doctors (separate from the study doctors) you see that you are participating in this research study.

If your anemia becomes severe while you are on study, then a transfusion may be recommended. If mucositis develops, the prohibited medicines can be allowed for treatment of the condition. If you experience an intolerable side effect while on study, you may be taken off study. If you leave the study early for any reason, your doctor will continue to follow your progress for 4 weeks and will access your medical records for a minimum of 1 year after the last dose of study drug (either palifermin or placebo) was given.

At your end of study visit, you will be evaluated for your disease status with imaging studies [computed tomography (CT) scans or magnetic resonance images (MRI)] and your weight and vitals signs will be measured. You will report any medications you have taken since your last visit and any side effects or blood transfusion that you have had. You will also have a final blood draw (about 3 teaspoons) for routine tests.

The total length of your involvement in this study is expected to be about 18 weeks (4 to 5 months).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with sarcoma which is locally advanced, at high risk for relapse or metastatic for whom treatment with high dose doxorubicin (90 mg/m2) with ifosfamide (AI) or cisplatinum (AP) is indicated.
2. Patients (male and female) with childbearing potential (defined as not post-menopausal for 12 months, negative blood pregnancy test, or no previous surgical sterilization) must use adequate birth control.
3. Adequate hematologic (Absolute neutrophil count (ANC)>/= 1500/mm^3, >/= Hgb 10gm/dL, platelet count >/= 150,000/mm^3), renal (serum creatinine </= 1.5mg/dL), hepatic (serum bilirubin count </= 1.5 * normal and SGPT < 3 * normal) functions.
4. Karnofsky Performance Status >/= 80.
5. Signed informed consent form.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Patients with comorbid condition which renders patients at high risk of treatment complication.
3. Patients with metastatic disease to CNS.
4. Patient has uncontrolled angina, congestive heart failure (New York Heart Association > class II or known ejection fraction < 40%), uncontrolled cardiac arrhythmia, acute myocardial infarction within 3 months or has uncontrolled hypertension.
5. Patient has an active seizure disorder. Patients with a previous history of seizure disorders will be eligible for the study, if they have had no evidence of seizure activity, and they have been free of antiseizure medication for the previous 5 years.
6. Prior surgery or radiotherapy (RT) within 2 weeks of study entry.
7. Prior treatment with palifermin, or other keratinocyte growth factors (eg, KGF-2).
8. Thirty days or less since receiving an investigational product or device in another clinical trial. Current enrollment in another clinical trial is not permitted unless the sole purpose of the trial is to obtain post-treatment data on the subject (eg, long-term follow-up or survival data).
9. Known sensitivity to any of the products to be administered during this study, including Escherichia coli-derived products.
10. Psychological, social, familial, or geographical reasons that would prevent scheduled visits and follow-up.
11. Patients with a history of pancreatitis.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2005-12; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saroj Vadhan-Raj, M.D., Principal Investigator — University of Texas MDAnderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Result] Vadhan-Raj S, Trent J, Patel S, Zhou X, Johnson MM, Araujo D, Ludwig JA, O'Roark S, Gillenwater AM, Bueso-Ramos C, El-Naggar AK, Benjamin RS. Single-dose palifermin prevents severe oral mucositis during multicycle chemotherapy in patients with cancer: a randomized trial. Ann Intern Med. 2010 Sep 21;153(6):358-67. doi: 10.7326/0003-4819-153-6-201009210-00003. PMID 20855800
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 12/2005 to 02/2008. All recruitment done at UT MD Anderson Cancer Center.
Pre-assignment Details: Of the 49 enrolled, one participant withdrew before assignment to groups.
Groups:
- Palifermin: Palifermin + Chemotherapy (AI or AP Regimen);
  AI = Doxorubicin (Adriamycin) + Ifosfamide:
  Palifermin 180 mcg/kg 3 days prior to chemotherapy; Adriamycin 30 mg/m^2 intravenous (IV) for 72 hours starting Days 0 for total 90 mg/m^2. Ifosfamide 2.5 g/m^2 IV bolus Days 0-3 (total 10 g/m^2); Vincristine 2 mg IV Day 0.
  AP=Doxorubicin (Adriamycin) + Cisplatin:
  Palifermin 180 mcg/kg 3 days prior to chemotherapy; Adriamycin 30 mg/m^2 IV continuous infusion for 72 hours starting Day 0(total = 90 mg/m^2); Cisplatin 120 mg/m^2 on day 0.
- Placebo: Placebo + Chemotherapy (AI or AP Regimen):
  AI = Doxorubicin (Adriamycin) + Ifosfamide:
  A single dose placebo 3 days prior to chemotherapy; Adriamycin 30 mg/m^2 intravenous (IV) for 72 hours starting Days 0 for total 90 mg/m^2. Ifosfamide 2.5 g/m^2 IV bolus Days 0-3 (total 10 g/m^2); Vincristine 2 mg IV Day 0.
  AP=Doxorubicin (Adriamycin) + Cisplatin:
  A single dose placebo 3 days prior to chemotherapy; Adriamycin 30 mg/m^2 IV continuous infusion for 72 hours starting Day 0(total = 90 mg/m^2); Cisplatin 120 mg/m^2 on day 0.
Period: Overall Study
Arm/Group | Palifermin | Placebo
Started | 32 | 16
Completed | 20 | 5
Not Completed | 12 | 11
Not completed — Disease progression | 4 | 2
Not completed — Chemotoxicity | 2 | 0
Not completed — Open-label palifermin | 2 | 7
Not completed — Surgery | 3 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Radiation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Palifermin | Placebo | Total
Number analyzed (Participants) | 32 | 16 | 48
Age, Customized [Median (Full Range); unit: years] | 42 [17 to 63] | 39 [15 to 64] | 42 [15 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 8 | 23
  Male | 17 | 8 | 25
Region of Enrollment [Number; unit: participants]
  United States | 32 | 16 | 48
Number of participants on two different chemotherapy regimens. [Number; unit: Participant] — Number of participants on two different chemotherapy regimens:AI; AP.
  Participant
    Number of participants on AI chemotherapy | 30 | 15 | 45
    Number of participants on AP chemotherapy | 2 | 1 | 3
Participants' Completion of 6 Blinded Cycles [Number; unit: participants] — Number of participants completing six (6) blinded treatment cycles; one cycle equals 3 weeks.
  participants
    Completed 6 Cycles | 20 | 5 | 25
    Not Completed 6 Cycles | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Incidence Rate of Oral Mucositis
Description: Cumulative incidence of World Health Organization (WHO) grade 2 or > mucositis (moderate to severe) in participants completing up to 6 blinded cycles. Rate defined as participants who had Grade 2 or > divided by total number of participants who completed up to 6 blinded cycles.
  WHO Criteria of Grade 1: possible buccal mucosal scalloping with/without erythema; No ulcers; swallows solid diet. Grade 2: ulcers with or without erythema; swallow solid diet. Grade 3: ulcers with/without (extensive) erythema; swallow liquid, not solid diet. Grade 4: mucositis to extent alimentation not possible.
Time Frame: Within 6 blinded cycles (3-week cycles), up to 18 weeks.
Population: Intention to treat (ITT).
Measure: Mean (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Palifermin | Placebo
Number analyzed (Participants) | 32 | 16
Percentage of Participants
  Cumulative incidence of WHO grade 2 or higher muco | 44 [24 to 62] | 88 [52 to 97]
  Cumulative Incidence of WHO Grade 3 or 4 Mucositis | 13 [4 to 27] | 51 [23 to 73]
Statistical Analysis 1: Comparison: Palifermin vs Placebo; Test type: Superiority or Other; p < 0.001, Fine and Gray method

2. Primary Outcome: Median Maximum Score for Patient Reported Outcomes in 2 Blinded Cycles
Description: Median maximum score (0 to 10, with 10 being the worst) for participant-reported outcomes in the first 2 blinded cycles for Mouth Pain, Overall Mouth and Throat Soreness, and Rectal Soreness while median maximum score for Swallowing, Drinking and Eating Difficulty (0 to 4, with 4 being the difficult).
Time Frame: Within the first 2 blinded cycles (3-week cycles), up to 6 weeks.
Population: Intention to treat (ITT).
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Palifermin | Placebo
Number analyzed (Participants) | 32 | 16
Units on a scale
  Mouth Pain | 1 [0 to 7] | 5 [0 to 10]
  Overall Mouth and Throat Soreness | 1 [0 to 9] | 5.5 [0 to 9]
  Rectal Soreness | 0 [0 to 9] | 4 [0 to 10]
  Drinking Difficulty | 0 [0 to 3] | 1.5 [0 to 3]
  Eating Difficulty | 0 [0 to 4] | 2 [0 to 4]
  Swallowing Difficulty | 0 [0 to 3] | 2 [0 to 4]

ADVERSE EVENTS:
Time Frame: 2 years and 3 months.
Description: Adverse events reported were found in the first two blinded cycles.
Arm/Group | Palifermin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/16
Other Adverse Events (participants affected / at risk) | 31/32 | 8/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Palifermin (N=32) | Placebo (N=16)
Increased thickness of oral mucosa (General disorders) | 30 | 5
Altered taste (General disorders) | 20 | 4
Flushing (General disorders) | 16 | 3
Film coating in mouth (General disorders) | 17 | 3
Increased sensitivity in tongue or gums (General disorders) | 15 | 2
Warm sensation (General disorders) | 11 | 0
Increased saliva (General disorders) | 8 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No